CLINICAL TRIAL: NCT04983810
Title: A Phase 1/2, Open-label, Multicenter Study to Investigate the Safety, Pharmacokinetics, and Efficacy of Fadraciclib (CYC065), an Oral CDK 2/9 Inhibitor, in Subjects With Advanced Solid Tumors and Lymphoma
Brief Title: A Study to Investigate Fadraciclib (CYC065), in Subjects With Advanced Solid Tumors and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYC065-101
Record Dates: First submitted 2021-07-12; First posted 2021-07-30 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult; Lymphoma
Keywords: Solid tumor; lymphoma
MeSH Terms: conditions — Lymphoma | interventions — CYC065

STUDY DESIGN:
Intervention Model Description: Dose escalation in Phase 1 part.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I Dose escalation (Experimental): Phase I = Fadraciclib administered orally in escalating doses starting at 50mg bid MWF for 3 weeks of a 4 week cycle. Subsequent cohorts will escalate in dose and schedule until optimized phase 2 dose and schedule is achieved.
  Phase 2 = Recommended Fadraciclib phase 2 dose and schedule administered orally in 28 day cycles.
  Interventions: Drug: Fadraciclib

INTERVENTIONS:
Drug: Fadraciclib — Fadraciclib is a highly selective, orally- and intravenously- available, 2nd generation amino-purine inhibitor of CDK2 and CDK9.
  Other Names: CYC065

SUMMARY:
This is a 2-part, phase 1/2, open-label, multicenter study designed to evaluate the safety, tolerability, PK, pharmacodynamics, PGx, and efficacy of fadraciclib administered orally BID. This study consists of Phase 1 and Phase 2 components in subjects with advanced solid tumors and lymphoma who have progressed despite having standard therapy or for which no standard therapy exists.

DETAILED DESCRIPTION:
Phase 1 part of the study will consist of a dose-escalation and a dose-finding component .

Phase 2 will enroll subjects with locally advanced, recurrent, or metastatic, histologically confirmed advanced solid tumors or lymphoma, who have failed all standard therapies or for whom standard therapy does not exist, into 8 groups:

Group 1: Endometrial or Ovarian cancer

Group 2: Biliary tract cancer

Group 3: HCC

Group 4: Breast cancer, meeting any of the following criteria:

* HER-2 refractory MBC
* HR positive, HER-2 negative, MBC post-CDK4/6 inhibitor
* Triple-negative breast cancer (TNBC)

Group 5: B-cell lymphoma

Group 6: T-cell lymphoma (CTCL and PTCL)

Group 7: mCRC, including KRAS mutated mCRC

Group 8: Basket cohort: Tumor types suspected to have a related mechanism of action such as MCL1, MYC or CCNE amplification/overexpression not included in previous groups.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years
2. Subjects with histological- or cytological-confirmed, advanced cancer who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists

   1. For Phase 1, all tumor types may be enrolled
   2. For Phase 2, subjects will be enrolled as per the study design section above
3. ECOG performance status of 0 or 1
4. Women of childbearing potential (WOCBP) must have a negative pregnancy test (urine or serum) within 7 days prior to starting the study drug. Both males and females must agree to use effective birth control during the study (prior to the first dose and for 6 months after the last dose) if conception is possible during this interval.
5. Subjects must be able to swallow and retain orally administered medication and not have any clinically significant GI abnormalities that may alter the absorption, such as malabsorption syndrome or major resection of the stomach or bowels.
6. Able to agree to and sign t he informed consent and to comply with the protocol.

Exclusion criteria

1. Subjects with a history of brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases. Subjects with treated brain metastases that are asymptomatic and have been clinically stable for at least 4 weeks will be eligible.
2. Subjects who have not received vaccines for SARS-COV-2 within last 3 months and have suspected signs and symptoms of COVID-19 or a recent history (within 14 days) of contact with any COVID-19 positive subject/isolation/quarantine or subjects with confirmed COVID-19.
3. Subjects with a history of another primary malignancy, other than:

   1. Carcinomas in situ, e.g., breast, cervix, and prostate
   2. Locally excised nonmelanoma skin cancer
   3. No evidence of disease from another primary cancer for 2 or more years and has not taken any anti-cancer treatment in 2 years.
4. Any other clinically significant acute or chronic medical or psychiatric condition or any laboratory abnormality that may increase the risk associated with study drug administration or may interfere with the interpretation of study results.
5. Diseases that significantly affect GI absorption of fadraciclib.
6. Subjects who have impaired cardiac function or clinically significant cardiac disease.
7. Presence of active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment
8. Presence of an active infection requiring intravenous antibiotics
9. Presence of known history of human immunodeficiency virus-1/2 with uncontrolled viral load and on medications that may interfere with metabolism
10. Presence of active hepatitis B virus (HBV) or hepatitis C virus (HCV).
11. Chemotherapy, biologic therapy, targeted therapy, immunotherapy, extended-field radiotherapy, or investigational agents within 5 half-lives or 3 weeks (whichever is shorter) prior to administration of first dose of study drug on Day 1 or have not recovered from the side effects of such therapy.
12. Major surgery/surgical therapy for any cause within 4 weeks of the first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 months
  The incidence rate of dose-limiting toxicities (first cycle only) at each dose level
Overall Response Rate (ORR) | 18 months
  Assessment of response criteria according to RESIST, Lugano or mSWAT

SECONDARY OUTCOMES:
Adverse events | 24 months
  Type, frequency, and severity of adverse drug reactions
AUC | 6 months
  Fadraciclib plasma concentrations
Cmax | 6 months
  Fadraciclib plasma concentrations
Tmax | 6 months
  Fadraciclib plasma concentrations
T1/2 | 6 months
  Fadraciclib plasma concentrations

OTHER OUTCOMES:
Pharmacodynamics | 6 months
  To investigate CDK9-dependent transcription inhibition as assessed by differential target gene expression relative to baseline.
Pharmacogenomics | 24 months
  To investigate plasma cell-free DNA mutation and copy number variation profile of fadraciclib as determined by NGS.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Kirschbaum, MD, Study Chair — Cyclacel Pharmaceuticals, Inc.
Locations (4):
- United States (2):
  - City of Hope, Duarte, California
  - MD Anderson Cancer Center, Houston, Texas
- Seoul National University Hospital, Seoul, South Korea
- Hospital Universitario Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No